CLINICAL TRIAL: NCT04829539
Title: Multicenter Randomized Controlled Trial Comparing Brief Behavioral Therapy for Cancer Related Insomnia (BBT-CI) and Healthy Eating Education Learning (HEAL)
Brief Title: Comparing Brief Behavioral Therapy (BBT-CI) and Healthy Eating Education Learning (HEAL) for Cancer-Related Sleep Problems While Receiving Cancer Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Mustian, Study Co-Chair, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: URCC-19185; NCI-2020-07175 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC19185 (Other: University of Rochester NCORP Research Base); URCC-19185 (Other: DCP); URCC-19185 (Other: CTEP); R01CA214647 (NIH); R01CA239714 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-04-02 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After completion of all baseline assessments, the coordinator will tell the study participant which group they are in but will not reveal which intervention is hypothesized to have a greater effect on insomnia. Both interventions will be presented with equipoise. The investigator and the statistical team will be blinded to the intervention group. The rest of the study staff will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (BBT-CI) (Experimental): Patients complete face to face/video sessions with a trained staff member. Patients also complete phone sessions.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (HEAL) (Active Comparator): Patients complete face to face/video sessions with a trained staff member. Patients also complete phone sessions.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive BBT-CI
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Group I (BBT-CI)
Behavioral: Behavioral Intervention — Receive HEAL
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Group II (HEAL)
Other: Electronic Health Record Review — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares BBT-CI to HEAL for the reduction of insomnia in patients with stage I-IV cancer who are receiving cancer treatment. Cancer treatment can cause side effects such as sleep problems. Sleep problems such as insomnia, are common for cancer patients. Insomnia can be described as difficulty falling asleep, waking up many times during the night or waking up earlier than patient would like. Insomnia can increase fatigue and worsen quality of life. This trial may help researchers determine which treatment works better in reducing insomnia, BBT-CI or HEAL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of BBT-CI compared to HEAL for treating insomnia as measured by the Insomnia Severity Index (ISI) at post-intervention.

SECONDARY OBJECTIVE:

I. Determine the efficacy of BBT-CI compared to HEAL for improving sleep efficiency as measured via actigraphy at post-intervention.

MECHANISTIC OBJECTIVE:

I. Examine the efficacy of BBT-CI compared to HEAL for regulating circadian rhythms as measured via actigraphy (i.e., Mesor, Acrophase, Amplitude, I<O dichotomy index).

EXPLORATORY OBJECTIVES:

I. Examine potential moderators of BBT-CI effects on insomnia (ISI). II. Examine potential mediators of BBT-CI effects on insomnia (ISI). III. Determine the efficacy of BBT-CI compared to HEAL for treating insomnia as measured by the Insomnia Severity Index at the 6-month follow-up.

IV. Determine the efficacy of BBT-CI compared to HEAL for improving sleep efficiency as measured via actigraphy at the 6-month follow-up.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (BBT-CI): Patients complete face to face/video sessions with a trained staff member. Patients also complete phone sessions.

GROUP II (HEAL): Patients complete face to face/video sessions with a trained staff member. Patients also complete phone sessions.

After completion of study, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Be diagnosed with cancer (stage I, II, III, or IV) with a life expectancy of at least 12 months
* Be currently receiving any cancer treatment (surgery alone is excluded)
* Report sleep disturbance of 3 or greater on the sleep disturbance question: "Rate your sleep disturbance in the past 2 weeks on a scale from 0-10, 0 is no problems and 10 is having the most severe problems"
* Have a score of 2, 1, or 0 on the Eastern Cooperative Oncology Group (ECOG) performance status scale
* Be able to speak, understand and read English to participate in the study assessments and interventions

Exclusion Criteria:

* Have a clinical diagnosis of obstructive sleep apnea or restless leg syndrome (even if controlled)
* Be engaged in a formal cognitive behavioral therapy for insomnia program presently or in the past 30 days. Use of sleep medications are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | post intervention
  Will evaluate the mean between arm difference in ISI score change from time point baseline to post-intervention. To assess this, will use analysis of covariance model with ISI at post-intervention as the outcome, study arm (group) as a fixed effect and baseline ISI as a covariate. Will test baseline group interaction.

SECONDARY OUTCOMES:
Sleep efficiency | post intervention
  Will be measured via actigraphy.
Circadian phenomena | Up to 6 months post intervention
  Circadian phenomena will be measured via actigraphy (Mesor, Acrophase, Amplitude, I < O dichotomy index).

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Palesh, PhD, Principal Investigator — Massey Cancer Center
Locations (153):
- United States (153):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Waverly Hematology Oncology, Cary, North Carolina
  - Outer Banks Hospital, Nags Head, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Valley Health / Winchester Medical Center, Winchester, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811